CLINICAL TRIAL: NCT00107029
Title: Evaluation of HIV-Specific CD8+ T-Cell Responses and Escape Mutations as Explanations for the Observed Differences in Disease Progression Conferred by HLA Class I Alleles
Brief Title: Evaluation of Genetic Markers as Explanations for the Observed Differences in Disease Progression in HIV+ Youth
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 026
Record Dates: First submitted 2005-04-04; First posted 2005-04-05 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infection
Keywords: HIV infection; CD8+ T-cells; HIV-1 genotype
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Biomedical HIV-1 related data and samples are available for the time the subjects were enrolled in REACH. HIV-1 genotyping will certainly be possible from these retrospective samples and the stored PBMCs will be evaluated for usefulness in the HIV-1 specific assays. Prospectively, samples will be collected every six months over a two-year period to evaluate both HIV-1 specific CD8+ T cell responses and the dominant HIV-1 genotype longitudinally.
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol is a study of HIV+ young people who were identified as having certain HIV-1 specific T-cell responses and genetic markers while previously enrolled in the 5-year longitudinal adolescent study, "REACH." Blood samples will be collected, a medical and medication history and physical examination will be performed every 6 months for a total of 2 years.

DETAILED DESCRIPTION:
Numerous studies have demonstrated an association between HLA class I genotypes with differing progression to AIDS in individuals who are followed after being off antiretroviral therapy. These studies do not always associate the same HLA class I alleles with the risks of HIV-1 disease progression; however they consistently demonstrated that HLA-B*35 and B*53 portend a bad outcome compared to the better outcome observed in HLA-B*27 and B*57 carriers. Despite this information, very little data exists to explain the mechanism of this association.

This longitudinal study will look at the HIV-1 specific CD8+ T-cell responses and the dominant HIV-1 genotype among individuals identified as HLA-B*27, B*35, B*53 and B*57 positive through studies done in collaboration with the REACH project.

ELIGIBILITY:
Inclusion Criteria:

* HLA-Class I HLA-B*27, B*35, B*53 and/or B*57 positive identified through the REACH study
* Subject's ability and willingness to provide written informed consent
* Subject's ability and willingness to be followed at least one year on this ATN 026 study

Exclusion Criteria:

* On chronic immunosuppressive therapy, not including topical or inhaled steroid use.
* Any prohibited medication listed in protocol within 2 weeks prior to the Entry visit labs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who were identified as HLA Class I HLA-B*27, B*35, B*53, and/or B*57 positive from the REACH study will be contacted for their interest in participating in this study. Only former REACH sites in the ATN will be eligible to enroll subjects into this study.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2002-12; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Demonstrate that few CTL escape mutations occur in HIV-1 specific CD8+ T cell epitopes that are HLA-B*27 and B*57 restricted, when compared to those restricted by HLA-B*35 and B*53. | 96 Weeks
  Demonstrate that few CTL escape mutations occur in HIV-1 specific CD8+ T cell epitopes that are HLA-B*27 and B*57 restricted, when compared to those restricted by HLA-B*35 and B*53.

SECONDARY OUTCOMES:
Demonstrate that CD8+ T cells have a high functional avidity to HLA-B*27 and B*57 bound epitopes when compared to those responding to HLA-B*35 and B*53 bound epitopes. | 96 Weeks
  Demonstrate that CD8+ T cells have a high functional avidity to HLA-B*27 and B*57 bound epitopes when compared to those responding to HLA-B*35 and B*53 bound epitopes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goepfert, MD, Study Chair — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami-Jackson Memorial Medical Center, Miami, Florida
  - Cook County Children's Hospital, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital at Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- See also: Website for the Adolescent Trials Network for HIV/AIDS Interventions — http://www.atnonline.org